CLINICAL TRIAL: NCT05474963
Title: Prospective Cohort Study of Sudden Sensorineural Hearing Loss in Wonju Severance Christian Hospital
Brief Title: Sudden Sensorineural Hearing Loss in Wonju Severance Christian Hospital
Status: Recruiting | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Tae Hoon Kong, MD, PhD, Assistant Professor, Wonju Severance Christian Hospital
Other Study IDs: WSCH-ENT-SSNHL-01
Record Dates: First submitted 2022-06-06; First posted 2022-07-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: SSNHL(Sudden Sensory Neural Hearing Loss); Sudden Hearing Loss; Hearing Loss, Idiopathic Sudden Sensorineural; Hearing Loss, Sudden
Keywords: Hearing Loss; Hearing Loss, sudden; SSNHL; Sudden sensorineural hearing loss; sudden sensory neural hearing loss
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SSNHL treated with WSCH protocol: SSNHL treated with WSCH protocol

SUMMARY:
This study is to build a cohort of sudden sensorineural hearing loss (SSNHL) patients. When the patient visited the Department of otolaryngology clinic for hearing loss, we can diagnose the SSNHL following the result of pure tone audiometry and the history of the patient. The cohort is a system that tracks the hearing recovery status, timing, and degree of recovery of patients who received cocktail therapy with or without high-dose steroids, vasodilators, antiviral agents, and intratympanic steroid injections, satellite ganglion block, and hyperbaric oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 20 years of age
* A patient who visited Wonju Severance Christian Hospital, Department of Otolaryngology and was diagnosed with sudden hearing loss as it was confirmed that hearing loss of 30dBHL or more occurred within 3 days at three consecutive frequencies in a pure tone audiometry test.
* Those who have fully explained the purpose and content of the study and voluntarily agreed to the written consent

Exclusion Criteria:

* If the patients do not want to or do not fill out the consent form
* If treatment is started for sudden hearing loss, but the possibility of other inner ear diseases including Meniere's disease is suspected due to repeated hearing loss, repeated recovery, dizziness, tinnitus, etc.
* Other cases where it is judged difficult to carry out the clinical trial due to the judgment of the person in charge of the above clinical trial

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the adults over 20yrs of age, diagnosed sudden sensorineural hearing loss at Wonju Severance Christian Hospital, Department of otolaryngology.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Hearing outcome 1 week - PTA | 1 week PTA
  Hearing change status near 1 weak after treatment start measured by pure tone audiometry1
Hearing outcome 3 weeks - PTA | 3 weeks PTA
  Hearing change status near 3 weaks after treatment start measured by pure tone audiometry
Hearing outcome 2 months - PTA | 2 month PTA
  Hearing change status near 3 weaks after treatment start measured by pure tone audiometry
Hearing outcome 3 months - PTA | 3 month PTA
  Hearing change status near 3 months after treatment start measured by pure tone audiometry
Hearing outcome 6 months - PTA | 6 months PTA
  Hearing change status near 6 months after treatment start measured by pure tone audiometry, which is final.

SECONDARY OUTCOMES:
Electrolytes and chemistries after high dose steroid therapy | 5 days electrolytes and chemistries
  The results of blood tests of electrolytes and chemistries at 5 days after treatment start.
  (Na, K, Cl, CO2, BUN, Cr, Glucose, Amylase, Total protein, Albumin, AST, ALT, ALP, r-GT, Total Bilirubin)

OTHER OUTCOMES:
Internal Acoustic canal MRI | MRI
  The baseline studies of internal acoustic canal MRI results of SSNHL patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chandrasekhar SS, Tsai Do BS, Schwartz SR, Bontempo LJ, Faucett EA, Finestone SA, Hollingsworth DB, Kelley DM, Kmucha ST, Moonis G, Poling GL, Roberts JK, Stachler RJ, Zeitler DM, Corrigan MD, Nnacheta LC, Satterfield L. Clinical Practice Guideline: Sudden Hearing Loss (Update). Otolaryngol Head Neck Surg. 2019 Aug;161(1_suppl):S1-S45. doi: 10.1177/0194599819859885. PMID 31369359
- [Background] Moon IS, Kim J, Lee SY, Choi HS, Lee WS. How long should the sudden hearing loss patients be followed after early steroid combination therapy? Eur Arch Otorhinolaryngol. 2009 Sep;266(9):1391-5. doi: 10.1007/s00405-009-0932-9. Epub 2009 Mar 13. PMID 19283405
- [Background] Moon IS, Lee JD, Kim J, Hong SJ, Lee WS. Intratympanic dexamethasone is an effective method as a salvage treatment in refractory sudden hearing loss. Otol Neurotol. 2011 Dec;32(9):1432-6. doi: 10.1097/MAO.0b013e318238fc43. PMID 22089956
- [Background] Rhee TM, Hwang D, Lee JS, Park J, Lee JM. Addition of Hyperbaric Oxygen Therapy vs Medical Therapy Alone for Idiopathic Sudden Sensorineural Hearing Loss: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2018 Dec 1;144(12):1153-1161. doi: 10.1001/jamaoto.2018.2133. PMID 30267033
- [Background] Park SM, Han C, Lee JW, Kong TH, Seo YJ. Does Herpes Virus Reactivation Affect Prognosis in Idiopathic Sudden Sensorineural Hearing Loss? Clin Exp Otorhinolaryngol. 2017 Mar;10(1):66-70. doi: 10.21053/ceo.2016.00360. Epub 2016 Jul 27. PMID 27459199